CLINICAL TRIAL: NCT06332508
Title: Pulsed Electromagnetic Fields (PEMFs) - A Highly Selective Breast CAncer Treatment pLatform (PASCAL), First-in-man Phase 1 Safety Trials
Brief Title: Pulsed Electromagnetic Fields (PEMFs) - A Highly Selective Breast CAncer Treatment pLatform (PASCAL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/00406
Record Dates: First submitted 2022-10-07; First posted 2024-03-27 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Pulsed Electromagnetic Fields (PEMFs)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEMFs prior to surgery (Experimental): During the study period, subjects will receive local magnetic therapy (PEMFs). The study aims to enrol subjects in 4 groups - in dose level 1 and 2 (subjects who do not need chemotherapy prior to surgery), PEMF will be administered prior to surgery;
  Interventions: Device: Pulsed electromagnetic fields (PEMFs)
- PEMFs prior to chemotherapy (Experimental): In dose level 3 and 4 (subjects who require chemotherapy), PEMF will be administered prior to chemotherapy.
  Interventions: Device: Pulsed electromagnetic fields (PEMFs); Drug: Anthracycline-based chemotherapy

INTERVENTIONS:
Device: Pulsed electromagnetic fields (PEMFs) — Device: PEMFs
  PEMFs treatment can be delivered up to 7 days prior to day of surgery (dose levels 1-2) or anthracycline-based chemotherapy (dose levels 3-4) to allow subject flexibility of timing and decrease the need for multiple visits. A research staff will be assigned to be with subject during the duration of PEMFs to monitor for any side effects during treatment.
Drug: Anthracycline-based chemotherapy — Drug: Anthracycline-based chemotherapy (doxorubicin, cyclophosphamide)
  At dose levels 3 and 4, two cohorts will be opened: the first cohort will undergo surgical resection immediately after completion of anthracycline-based chemotherapy, and the second cohort will undergo taxane-based chemotherapy following completion of anthracycline-based chemotherapy.
  Arms: PEMFs prior to chemotherapy

SUMMARY:
To assess the safety and tolerability of combined PEMFs and anthracycline-based chemotherapy in subjects who are undergoing neoadjuvant chemotherapy for breast cancer treatment.

DETAILED DESCRIPTION:
This is a single-center phase Ib study to investigate the safety and tolerability of the combination of PEMF with anthracycline-based chemotherapy. Subjects will be enrolled on a 3+3 dose escalation design from dose level 1 with a target to reach dose level 4, where PEMF can be administered prior to each cycle of anthracycline-based chemotherapy. In the first 2 dose levels, PEMFs will first be administered to subjects who are planned for upfront surgical resection to ensure that PEMFs is safe and tolerable for up to 0.5-hour. Once the duration of each PEMF treatment is established, PEMFs will then be added to anthracycline-based chemotherapy to investigate the safety and tolerability of the combination treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed breast carcinoma of any subtype (any estrogen receptor, progesterone receptor and HER2 receptor status)
2. ECOG 0-1.
3. Non-metastatic disease for which surgery of curative intent is planned upfront or after completion of neoadjuvant chemotherapy
4. Adequate organ function including the following:

   1. Bone marrow:

      1. Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 10^9/L
      2. Platelets >= 100 x 10^9/L
      3. Hemoglobin >= 8 x 10^9/L
   2. Hepatic:

      1. Bilirubin <= 1.5 x upper limit of normal (ULN),
      2. ALT or AST <= 2.5x ULN, (or <=5 X with liver metastases)
   3. Renal:

      1. Creatinine <= 1.5x ULN
5. Signed informed consent from subject or legal representative.
6. Able to comply with study-related procedures.

Exclusion Criteria:

1. Pregnancy.
2. Breast feeding.
3. Presence of fungating breast tumor or open wound in breast planned for PEMF.
4. Active bleeding disorder or bleeding site.
5. Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
6. Major surgery within 28 days prior to study administration.
7. Non-healing wound.
8. Active infection that in the opinion of the investigator would compromise the subject's ability to tolerate therapy.
9. History of significant neurological or mental disorder, including seizures or dementia.
10. Serious concomitant disorders that would compromise the safety of the subject or compromise the subject's ability to complete the study, at the discretion of the investigator.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer study - 99.9% breast cancer subjects are female. Male breast cancer is extremely rare and thus males will not be recruited
Enrollment: 36 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE 5.0 | up to 6 months
  Toxicity to treatment as assessed by Common Terminology Criteria for Adverse Events 5.0. Grade 1-5 refer to the severity of the adverse event with higher grade indicating greater severity. Grade 3 and above will be considered severe.
  A dose limiting toxicity will be defined as Grade 3 or above toxicity of the following:
  a) pain in breast where PEMF was applied
  * Increased intra-operatively bleeding whereby surgical bed require a longer period of hemostases
  * Post-surgical complications including delay wound healing (open wound of more than 5 days post-surgery), wound infection and wound dehiscence, hematoma formation

SECONDARY OUTCOMES:
Treatment response as assessed by clinical measurement of tumor size using calipers | up to 6 months
  Subjects should have documented the size of the tumor through clinical measurement using calipers at each assessment visit. Wherever possible, documentation of radiological size based on mammogram, ultrasound or magnetic resonance imaging should also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Wong, Medical Degree, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tai YK, Chan KKW, Fong CHH, Ramanan S, Yap JLY, Yin JN, Yip YS, Tan WR, Koh APF, Tan NS, Chan CW, Huang RYJ, Li JZ, Frohlich J, Franco-Obregon A. Modulated TRPC1 Expression Predicts Sensitivity of Breast Cancer to Doxorubicin and Magnetic Field Therapy: Segue Towards a Precision Medicine Approach. Front Oncol. 2022 Jan 24;11:783803. doi: 10.3389/fonc.2021.783803. eCollection 2021. PMID 35141145
- [Background] Haidinger R, Bauerfeind I. Long-Term Side Effects of Adjuvant Therapy in Primary Breast Cancer Patients: Results of a Web-Based Survey. Breast Care (Basel). 2019 Apr;14(2):111-116. doi: 10.1159/000497233. Epub 2019 Feb 15. PMID 31798383